CLINICAL TRIAL: NCT07038239
Title: Deciphering MORC2 Genotype/Phenotype Correlation to Improve Patient Diagnostic
Brief Title: Genotype/Phenotype Correlation of MORC2 Mutations
Acronym: PhenoMORC2
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0647; 2025-A00225-44 (Other: N° ID-RCB)
Record Dates: First submitted 2025-05-27; First posted 2025-06-26 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Charcot Marie Tooth Disease; DIFGAN; Developmental Delay (Disorder); Impaired Growth; Dysmorphic Facies and Axonal Neuropathy
Keywords: Charcot-Marie-Tooth; DIFGAN; Human silencing hub complex; genotype-phenotype correlation; MORC2; DNA dalage repair; transcriptional modulation; EPIGENETIC
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Developmental Disabilities | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Charcot-Marie-Tooth patients : Patients presenting with length-dependent sensitive-motor axonal neur: Patients presenting with length-dependent sensitive-motor axonal neuropathy
  Interventions: Diagnostic Test: Skin biopsy; Diagnostic Test: Blood sample
- DIFGAN patients: Patients presenting with DIFGAN syndrome : developmental delay, impaired growth, dysmorphic facies and axonal neuropathy
  Interventions: Diagnostic Test: Skin biopsy; Diagnostic Test: Blood sample
- Control: Control group without any neurological disorder

INTERVENTIONS:
Diagnostic Test: Skin biopsy — under the arm using a 3 mm punch, with local anaesthesia, in the investigating centres.
  Groups: Charcot-Marie-Tooth patients : Patients presenting with length-dependent sensitive-motor axonal neur; DIFGAN patients
Diagnostic Test: Blood sample — 3 classical 4ml tubes samples per patients, using the routine blood sampling technique, in the investigating centres.
  For children, blood sampling volume will be adapted to the patient's weight according to L.1121-1 of the French public health code.
  Groups: Charcot-Marie-Tooth patients : Patients presenting with length-dependent sensitive-motor axonal neur; DIFGAN patients

SUMMARY:
The Microrchidia CW-type zinc finger 2 (MORC2) gene encodes a protein expressed in all tissues and enriched in the brain. It is involved in Charcot-Marie-Tooth disease, with mire than 30 families presenting MORC2 mutations. Recently, MORC2 mutation have been shown to be responsible for more complex phenotypes like DIFGAN: developmental delay, impaired growth, dysmorphic facies and axonal neuropathy.

Different mutations are responsible from a diverse spectrum of phenotype, from CMT to DIFGAN.

MORC2 is involved, through its ATPase activity, in DNA repair, chromatin remodeling and epigenetic silencing via the Human silencing hub (HUSH) complex. Our hypothesis is that the hypo- or hyper-activation of the HUSH complex by different MORC2 mutations could be responsible for different phenotypes in patients. The aim of this study is to perform a genotype-phenotype correlation study in patients presenting MORC2 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a mutation in the MORC2 gene, identified during an evaluation for peripheral neuropathy or intellectual disability
* Patient has undergone electromyography (EMG) or is able to undergo EMG during the inclusion visit
* Affiliation with the national health insurance system
* Informed consent from the patient if an adult, or from parents/legal guardians if the patient is a minor

Exclusion Criteria:

* Presence of another mutation responsible for peripheral neuropathy or intellectual disability
* Refusal to undergo biological sample collection
* Regulatory exclusion criteria:
* Pregnant, postpartum, or breastfeeding women
* Individuals deprived of liberty by judicial or administrative decision
* Individuals not affiliated with a social security system or not benefiting from an equivalent health coverage scheme

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will focus on children and adults suffering from a MORC2 gene mutation, and presenting a CMT or DIFGAN phenotype.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Epigenetic biomarker levels | At inclusion
  Quantification of epigenetic biomarkers in patient and control-derived cells (number of reads in patients vs controls)

SECONDARY OUTCOMES:
RNA-seq | At inclusion
  quantification of specific mRNA sequences in patient-derived cells (RNA copy number in patient vs control)
Detection and quantification of specific nucleic acid biomarkers in patient's serum | At inclusion
  Quantification of nucleic acid biomarkers in the patient's serum (number of reads in patients vs control)
Quantification of nucleic acid biomarkers in patient's cerebrospinal fluid | At inclusion
  Quantification of nucleic acid biomarkers in the patient's cerebrospinal fluid (CSF) (number of reads in patients vs control)
Quantification of proteic biomarkers in patient's serum | At inclusion
  Quantification of proteic biomarkers in the patient's serum (µg/mL)
Quantification of proteic biomarkers in patient's cerebrospinal fluid (CSF) | At inclusion
  Quantification of proteic biomarkers in the patient's cerebrospinal fluid (CSF)(µg/mL)

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU de Besançon, Besançon
  - CHRU Brest, Brest
  - CHU Grenoble, Grenoble
  - CH de Versailles, Le Chesnay
  - Service de Génétique moléculaire, pharmacogénétique, hormologie Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hospices Civils de Lyon, Lyon
  - CHU Marseille, Marseille
  - CHU de Nantes, Nantes
  - CH Pitié Salpêtrière, Paris
  - Hôpital Necker, Paris
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No